CLINICAL TRIAL: NCT01378247
Title: Family Focused Nursing for Outpatients With Heart Failure
Brief Title: Multicenter Study of Family Nursing to Treat Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Vejle Hospital (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Birte Oestergaard, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UNR-20110068-3
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Family Nursing; Health-Related Quality of Life; Heart Failure Clinic
MeSH Terms: conditions — Heart Failure | interventions — Nursing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Pharmacological treatment, patient information and counselling according to international and national guidelines by health professionals specialized in heart failure.
- Family Focused Nursing (Experimental): Family Focused Nursing and treatment as usual
  Interventions: Behavioral: Family Focused Nursing

INTERVENTIONS:
Behavioral: Family Focused Nursing — All patients receive treatment as usual. Additionally, patients in the intervention arm receives family focused nursing consultations which are structured as outpatient sessions focusing on change, improvement and/or maintenance of family function within cognitive, affective and behavioral knowledge. Each session is organized and individualized according to the wishes and needs for education and counseling of the families within a period of six months.
  Other Names: Family; Nursing; Heart Failure
  Arms: Family Focused Nursing

SUMMARY:
The purpose of this study is to determine whether Family Focused Nursing are effective in the treatment of heart failure outpatients with respect to health-related quality of life.

DETAILED DESCRIPTION:
Quality of life is impaired among patients with heart failure and their next of kin compared to other patients with chronic diseases. Besides, there are still a number of patients who misunderstand or have difficulties remembering the counseling they are provided during the course of illness. International guidelines recommend that the patient's relatives are involved in patient education as well as the treatment. Family interventions might contribute to improvement in quality of life, enhanced illness-management and delayed readmission and mortality among patients with heart failure. However, up till today, only two observational studies have investigated the effect of family intervention on outcomes of treatment for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Referred to follow-up nursing treatment in nurse-led heart failure clinic
* Diagnosed chronic heart failure, based on systolic dysfunction (left ventricular ejection fraction (LVEF) ≤40%)
* New York Heart Association (NYHA) classification II-IV symptoms
* Signed informed consent

Exclusion Criteria:

* Patients not understanding or talking danish
* In terminal phase of another serious illness such as i.e. cancer with expected lifetime less than 6 months
* Patients not giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life assessed by ≥6 point in Kansas City Cardiomyopathy Questionnaire summary score | Baseline, three, six and twelve months
  The effect of intervention on primary outcome are investigated as longitudinal data at three, six and twelve month. The data are analysed using mixed models

SECONDARY OUTCOMES:
Change in European Heart Failure Self-Care Behavior Scale | Baseline, three, six and twelve months months
Change in Family Functioning, Health and Social Support scale | Baseline, three, six and tvelve months
Change in Self-Efficacy for Managing Chronic Disease 6-item scale | Baseline, three, six and tvelve months
Change in Major Depression Inventory diagnostic scale | Baseline, three, six and tvelve months
Time for the emergence of total re-admission and re-admission for heart failure | One year
Time for the emergence of mortality | One year

CONTACTS AND LOCATIONS:
Overall Officials: Birte Oestergaard, PhD, Principal Investigator — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Data will be entered into Odense Patient data Explorative Network (OPEN) database